CLINICAL TRIAL: NCT06900478
Title: Icariin Soft Capsules Combined With TACE as Adjuvant Therapy for Hepatocellular Carcinoma With High-Risk Recurrence Factors:A Single-Center, Prospective Study
Brief Title: Icariin Soft Capsules Combined With TACE as Adjuvant Therapy for HCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hua Li (Other)
Responsible Party: Sponsor-Investigator, Hua Li, Director, Liver Surgery and Liver Transplantation Center, Third Affiliated Hospital, Sun Yat-Sen University
Organization: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-349-02
Record Dates: First submitted 2025-03-20; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Hepatocarcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Icariin Soft Capsules + TACE (Experimental): TACE treatment was performed one month after surgery, and Icariin Soft Capsules for disease progression or study termination.
  Interventions: Drug: Icariin Soft Capsules+TACE

INTERVENTIONS:
Drug: Icariin Soft Capsules+TACE — TACE: perform preoperative infusion chemotherapy, then selectively inject 2 to 5 mL of iodized oil and embolize.
  Icariin Soft Capsules：take 6 tablets each time, orally, twice a day.

SUMMARY:
This is a prospective, single-center, phase II study，to evaluate the efficacy and safety of icariin soft capsules combined with TACE as adjuvant therapy in hepatocellular carcinoma (HCC) patients at high risk of recurrence after resection.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years;
* ECOG Performance Status (PS) of 0 or 1;
* Histologically or cytologically diagnosed as HCC
* Fully recovered from surgical resection or ablation prior to enrollment;
* Presence of the following high-risk recurrence factors after resection or ablation: tumor maximum diameter > 5 cm; multiple tumors; microvascular or major vascular invasion; margin distance from the tumor edge < 1 cm; poorly differentiated tumors (Edmondson grade III-IV); lymph node metastasis; persistent abnormal AFP or abnormal prothrombin (DCP);
* Child-Pugh class A5-B7;
* Expected survival time > 3 months;
* Normal major organ function: Hemoglobin ≥ 80 g/L, Absolute Neutrophil Count (ANC) ≥ 1.5 × 10^9/L, Platelet count ≥ 50 × 10^9/L, Serum albumin ≥ 30 g/L, Total bilirubin ≤ 2 ULN, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) ≤ 2.5 × ULN, Alkaline Phosphatase (ALP) ≤ 2.5 × ULN, Creatinine ≤ 1.5 × ULN and creatinine clearance ≥ 50 ml/min, International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 × ULN, Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN;
* Negative HIV test results at screening;
* Hepatitis B virus (HBV) DNA<500 IU/mL;
* No major vascular invasion (Vp3 or Vp4) of the portal vein or any level of major vascular invasion of the hepatic veins or inferior vena cava;
* Within 7 days prior to screening, women of childbearing potential must confirm a negative serum pregnancy test and agree to use effective contraception during the study drug administration and for 60 days after the last dose of the study drug;

Exclusion Criteria:

* Known cases of fibrolamellar hepatocellular carcinoma (HCC), sarcomatoid HCC, or mixed cholangiocarcinoma and HCC;
* HCC recurrence prior to study enrollment;
* Co-infection with HBV and delta hepatitis virus;
* Clinically significant ascites (Note: ascites detectable only through imaging studies are permitted to participate in the study);
* History of hepatic encephalopathy;
* Receipt of any other investigational drug treatment within 4 weeks prior to Day

  1 of Cycle 1;
* Presence of abdominal wall fistula, gastrointestinal perforation, refractory non-healing gastric ulcers, or history of active gastrointestinal bleeding within 6 months prior to enrollment;
* History of another malignancy tumor , except for the cured skin basal cell carcinoma and cervical carcinoma in situ)
* Active tuberculosis;
* Functional impairment of major organs (heart, lungs, kidneys, etc.), severe infections, or > grade 2 adverse events (Common Terminology Criteria for Adverse Events (CTCAE) version 5.0);
* Very early-stage HCC, solitary tumors, size < 2 centimeters;
* Any allergy to the drugs used in the TACE regimen or known components of epimedium soft capsules;
* History of organ transplantation;
* Pregnant or breastfeeding female patients, or those unwilling to use contraception during the trial;
* Any other diseases, metabolic disorders, abnormal physical examination results, or laboratory test results that raise suspicion of contraindications for the investigational drug, may affect the reliability of study results, or place the patient at high risk for treatment complications, or affect patient compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free Survival Rate | 12 months
  The proportion of patients who did not experience recurrence or death

SECONDARY OUTCOMES:
Disease Free Survival | 24 months
  DFS defined as the time from date of treatment until the date of recurrence or death due to any cause
Overall survival (OS) | 24 months
  OS defined as the time from date of treatment until the date of death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No